CLINICAL TRIAL: NCT05660356
Title: Growth Hormone Deficiency in Patients With Persistent Symptoms Following Concussion
Brief Title: Growth Hormone Deficiency in Mild Traumatic Brain Injury
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Chantel T Debert, Academic Physiatrist, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB22-1684
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Growth Hormone Treatment; Growth Hormone Deficiency; Concussion, Mild; Concussion Post Syndrome
Keywords: Growth Hormone Deficiency; Persistent Post-concussion Symptoms; Growth Hormone Therapy; Clinical Trial
MeSH Terms: conditions — Dwarfism, Pituitary; Brain Concussion; Post-Concussion Syndrome | interventions — Growth Hormone

STUDY DESIGN:
Intervention Model Description: Treatment group and placebo group. Participants assigned placebo group will be given the option to complete...
Who Masked: Participant
Masking Description: Participants will be masked to their assigned group. Following completion of the study, participants will be informed of their group allocation and be given the option to complete the treatment group if they were originally assigned to the placebo group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Growth Hormone (Experimental): Participants will perform daily at-home subcutaneous GH injections after receiving thorough at-home education training provided by a pharmaceutical nurse before and research personnel. The GH will be provided be Pfizer. Starting doses will be 0.2 ug/L and 0.3 ug/L for women taking exogenous oral estrogen.
  Interventions: Drug: Growth Hormone
- Placebo (Placebo Comparator): Participants will perform daily at-home subcutaneous placebo injections after receiving thorough at-home education training provided by a pharmaceutical nurse before and research personnel. Starting doses will be 0.2 ug/L and 0.3 ug/L for women taking exogenous oral estrogen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Growth Hormone — Pfizer provided GH therapy
  Other Names: Growth Hormone Therapy
  Arms: Growth Hormone
Drug: Placebo — Pfizer provided placebo
  Other Names: Placebo (no active therapy)
  Arms: Placebo

SUMMARY:
The goal of this randomized control trial is to test if growth hormone therapy is a safe and effective treatment for patients suffering from growth hormone deficiency and persistent post-concussion symptoms. The main questions it aims to answer are:

1. Is growth hormone therapy effective at mitigating persisting post-concussion symptoms in patients with growth hormone deficiency?
2. Is it feasible to conduct a larger trial to examine efficacy of growth hormone therapy in patients with persistent post-concussion symptoms and growth hormone deficiency?

Participants will be asked to complete an initial assessment for study inclusion and to complete clinical outcome questionnaires. If a participant meets study criteria they will be randomized to receive either growth hormone therapy (provided by Pfizer) or a placebo (provided by Pfizer). Participants will be instructed on how to self-administer their assigned drug daily for three months. Monthly follow-up visits will include a blood draw to measure a biomarker and clinical outcome questionnaires. At the final follow-up visit after three months, participants will learn what group they were assigned and given the option to complete the growth hormone therapy if they were originally assigned to the placebo group.

Researchers will compare the growth hormone therapy group to the placebo group to identify any potential differences in outcomes.

DETAILED DESCRIPTION:
Annually, over 250,000 Canadians and over 40 million individuals worldwide will suffer an uncomplicated concussion (head injury with no intracranial abnormalities seen on imaging). Most individuals will recover within weeks of injury but over 30% will have persistent profound symptoms (PPCS) that impedes daily function, work and social activities. To date, there are few evidence-based treatments available for patients suffering PPCS leaving patients and clinicians grasping for answers to improve health. The culminative numbers of Canadians that are living with PPCS following a concussion are staggering and symptoms impact individual's ability to work and actively contribute to society, increasing demands on health care resources, draining public supports and diminishing contribution to the national workforce. To date, there are no recommended evidence-based treatments available to improve PPCS. Current PPCS treatments are extrapolated from other conditions and often include trial and error. Hypopituitarism has been studied extensively in patients with more severe traumatic brain injuries (TBI), with growth hormone deficiency (GHD) being the most common hormone abnormality. Previous studies have examined GHD in patients with TBI due to complicated mild (evidence of intercranial abnormalities on imaging), moderate and severe TBI, but never uncomplicated mTBI (no intercranial abnormality on imaging) or concussion (terms used interchangeably in this document). These studies have shown GH therapy can significantly improve symptoms and function in patients with TBI often allowing them to return to previous work and social activities. Recent retrospective studies completed by CTD and collaborators found approximately 35-41% of patients with concussion referred for GH testing were GHD and 78% had a significant improvement in symptoms at 3 months post-treatment1. Treatment with GH provided significant improvement in symptoms, often allowing them to return to productive jobs, caregiver activities, leisure activities and greatly improving overall quality of life. This research project is incredibly important and novel as it will be the first study to prospectively follow patients with persistent symptoms following concussion to determine prevalence of growth hormone deficiency (GHD) and implement a randomized double blinded placebo controlled cross-over trial to explore the response to GH therapy.

A randomized double-blinded placebo control cross-over trial will be completed to determine efficacy of GH treatment in this population as well as feasibility of a larger trial. We will recruit 20 individuals for this pilot study. Inclusion criteria will include 1) persistent symptoms 6-months following concussion and 2) Peak GH of < 3 mcg/L following glucagon stimulation test (GST). We will exclude patients with other untreated pituitary hormone deficits (gonadotrophin, TSH, ACTH, diabetes insipidus).

We will perform a pilot trial in order to (1) determine GH therapy efficacy in patients with concussion and GHD and (2) assess the feasibility of a larger prospective study of this nature. We will collect demographic information, injury characteristics, symptom questionnaires, and results from GST and other endocrine testing. Primary outcome will include improvement on the QoL-AGHDA questionnaire (a quality of life questionnaire that has been validated in individuals with GHD) from baseline to 3 months following therapy. Secondary assessments will include cognition (RBANS - repeatable battery for the assessment of neuropsychological status), depression (PHQ9), anxiety (GAD7) and rivermead post-concussion symptom questionnaire (RPQ) pre-treatment and 3 months post-treatment. A Clinical follow-up and IGF-1 levels will be performed at 1 month intervals. Unblinding will occur at 3 months, and patients in the placebo group will have the opportunity to cross-over to the treatment group if they choose. Patients that cross over will complete an additional QoL-AGHDA questionnaire after three months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a concussion according to the American Congress of Rehabilitation Medicine criteria with persistent symptoms 6-months following concussion
* Peak growth hormone of < 3 mcg/L following glucagon stimulation test

Exclusion Criteria:

* Untreated pituitary dysfunction
* Moderate/severe TBI
* Intracranial abnormalities
* Chronic neurologic conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Baseline QoL-AGHDA | Minimum 6-months following injury (no maximum)
  Adult Growth Hormone Deficiency Assessment Quality of Life Questionnaire. A high score indicates a lower quality of life.
3-months QoL-AGHDA | 3-months after baseline
  Adult Growth Hormone Deficiency Assessment Quality of Life Questionnaire. A high score indicates a lower quality of life.

SECONDARY OUTCOMES:
Baseline RBANS | Minimum 6-months following injury (no maximum)
  Repeatable Battery for the Assessment of Neuropsychological Status. A higher score indicates better outcomes.
3-months RBANS | 3-months after baseline
  Repeatable Battery for the Assessment of Neuropsychological Status. A higher score indicates better outcomes.
Baseline GAD-7 | Minimum 6-months following injury (no maximum)
  General Anxiety Disorder 7. A higher score indicates worse outcomes.
3-months GAD-7 | 3-months after baseline
  General Anxiety Disorder 7. A higher score indicates worse outcomes.
Baseline PHQ-9 | Minimum 6-months following injury (no maximum)
  Personal Health Questionnaire 9. A higher score indicates worse outcomes.
3-months PHQ-9 | 3-months after baseline
  Personal Health Questionnaire 9. A higher score indicates worse outcomes.
Baseline RPQ | Minimum 6-months following injury (no maximum)
  Rivermead Post-Concussion Symptom Questionnaire. A higher score indicates worse outcomes.
3-months RPQ | 3-months after baseline
  Rivermead Post-Concussion Symptom Questionnaire. A higher score indicates worse outcomes.
Baseline QoLIBRI | Minimum 6-months following injury (no maximum)
  Quality of Life after Brain Injury. A higher score indicates better outcomes.
3-months QoLIBRI | 3-months after baseline
  Quality of Life after Brain Injury. A higher score indicates better outcomes.
Baseline Sleep and Concussion Questionnaire | Minimum 6-months following injury (no maximum)
  Sleep and Concussion Questionnaire. A higher score indicates worse outcomes.
3-months Sleep and Concussion Questionnaire | 3-months after baseline
  Sleep and Concussion Questionnaire. A higher score indicates worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Chantel T Debert, MD, MSc, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mercier LJ, Kruger N, Le QB, Fung TS, Kline GA, Debert CT. Growth hormone deficiency testing and treatment following mild traumatic brain injury. Sci Rep. 2021 Apr 20;11(1):8534. doi: 10.1038/s41598-021-87385-7. PMID 33879807